CLINICAL TRIAL: NCT00706888
Title: Study on Effects of a Dairy Product Based on Polyphenols and Enriched With Vitamins B6, B9 and B12 on Some Cardiovascular Factor of Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elvir SAS (Industry)
Collaborators: BioFortis (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Etude 9108
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Cardiovascular Risk Factors
Keywords: Reduction of cardiovascular factor of risk
MeSH Terms: interventions — Vitamin B 12; Polyphenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- 1 (Active Comparator): Female with active product
  Interventions: Dietary Supplement: Vitamins B6, B9 and B12 and polyphenols
- 2 (Active Comparator): Male with active product
  Interventions: Dietary Supplement: Vitamins B6, B9 and B12 and polyphenols
- 3 (Placebo Comparator): Female with placebo
  Interventions: Dietary Supplement: placebo
- 4 (Placebo Comparator): Male with placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Vitamins B6, B9 and B12 and polyphenols
  Arms: 1; 2
Dietary Supplement: placebo
  Arms: 3; 4

SUMMARY:
We put forward that polyphenols and vitamins have a cardiovascular prevention effect for subject with cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* BMI less than 33 kg/m²
* Waist measurement higher than 90 cm for woman and 100 cm for man
* Normal or controled blood pressure (less than 16/9)
* non-smoker
* Female with contraception

Exclusion Criteria:

* Food allergy
* Cardiovascular pathology
* Medical treatment for cholesterol
* Higher consumption for dairy product and red fruit

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Nantes, France